CLINICAL TRIAL: NCT06449651
Title: Double-blind, Randomized, Placebo-controlled Study Evaluating the Safety and Efficacy of Nipocalimab in Reducing the Risk of Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT) in At-risk Pregnancies
Brief Title: A Study of Nipocalimab in Reducing the Risk of Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT)
Acronym: FREESIA-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 80202135FNAIT3001; 80202135FNAIT3001 (Other: Janssen Research & Development, LLC); 2023-504307-88-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thrombocytopenia, Neonatal Alloimmune
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nipocalimab (Active Comparator): Maternal participants will receive nipocalimab Intravenously (IV).
  Interventions: Drug: Nipocalimab
- Placebo (Placebo Comparator): Maternal participants will receive placebo IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered intravenously.
  Other Names: JNJ-80202135; JNJ-86507083
  Arms: Nipocalimab
Drug: Placebo — Placebo will be administered intravenously.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of nipocalimab compared with placebo in reducing the risk of severe fetal and neonatal alloimmune thrombocytopenia (FNAIT).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and an estimated gestational age (GA; based on ultrasound dating) from Week 13 to 18 at randomization
* Has a history of greater than or equal to (>=) 1 prior pregnancy with fetal and neonatal alloimmune thrombocytopenia (FNAIT) (including neonatal platelet count less than (<) 150×10^9/Liter) with none of them affected by fetal/neonatal intracranial hemorrhage (ICH) or severe hemorrhage based on medical records
* Current pregnancy with presence of maternal anti- human platelet antigen (HPA)-1a alloantibody and positive fetal HPA-1a genotype as confirmed by cell-free fetal deoxyribonucleic acid (DNA) in maternal blood
* Health status considered stable by the investigator based on physical examination, medical history, vital signs, 12-lead Electrocardiogram (ECG), and clinical laboratory tests performed at screening
* For maternal participant and neonate/infant, willing to forego participation in another clinical study of an investigational therapy until the last follow-up visit

Exclusion Criteria:

* Currently pregnant with multiple gestations (twins or more)
* History of severe preeclampsia in a previous pregnancy
* History of myocardial infarction, unstable ischemic heart disease, or stroke
* Known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients (refer to the Investigator Brochure (IB))
* Has any confirmed or suspected clinical immunodeficiency syndrome or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2029-12-05 (Estimated); Study Completion 2029-12-11 (Estimated)

PRIMARY OUTCOMES:
Fetus/Neonate with Outcome of Death or Adjudicated Severe Bleeding or Platelet Count Less Than (<) 30*10^9/L | Up to 1 week post birth
  Outcome of fetus/neonate death or adjudicated severe bleeding up to the first week post birth or platelet count <30*10^9/L will be reported.

SECONDARY OUTCOMES:
Neonate/Fetus With Adjudicated Bleeding | Up to 1 Week post birth
  Neonate/fetus With adjudicated bleeding will be reported.
Platelet Count at Birth in a Neonate | At birth
  Platelet count at birth in a neonate will be reported.
Neonate/Fetus with Outcome of Death | Up to 1 Week post birth
  Fetus/neonate with outcome of death will be reported.
Platelet Count at Birth <10×10^9/L in a Neonate | At birth
  Platelet count at birth <10×10^9/L in a neonate will be reported.
Platelet Count at Birth <30×10^9/ L In a Neonate | At birth
  Platelet count at birth <30×10^9/L in a neonate will be reported.
Platelet Count at Birth <50×10^9/L In a Neonate | At birth
  Platelet count at birth <50×10^9/L in a neonate will be reported.
Platelet Count at Birth <150×10^9/L In a Neonate | At birth
  Platelet count at birth <150×10^9/L in a neonate will be reported.
Nadir Platelet Count of a Neonate Over the First Week Post Birth | Upto 1 Week post birth
  Nadir platelet count in a neonate will be reported.
Neonate/Fetus Requiring Platelet Transfusion(s) | Up to 1 Week post birth
  Neonate(s) who require at least one platelet transfusion(s) will be reported.
Number of Platelet Transfusion(s) in Neonate/Fetus | Up to 1 Week post birth
  Number of Platelet transfusion(s) per neonate will be reported.
Number of Donor Exposures for Platelet Transfusion(s) in Neonate/Fetus | Up to 1 Week post birth
  Number of donor exposures for neonates who received platelet transfusion(s) will be reported.
Neonate/Fetus With Adjudicated Severe Bleeding | Up to 1 week post birth
  Neonate/Fetus With adjudicated severe bleeding will be reported.
Neonates With Postnatal Intravenous Immunoglobulin (IVIG) for The Treatment of Thrombocytopenia | Up to 1 Week post birth
  Neonates with IVIG for the treatment of thrombocytopenia will be reported.
Maternal Participants With Treatment-Emergent Adverse Event (TEAE) | From randomization up to 24 weeks postpartum
  Maternal participants with a TEAE will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Maternal Participants With Serious Adverse Event (SAE) | From randomization up to 24 weeks postpartum
  Maternal participants with SAE will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. SAE is any untoward medical occurrence that at any dose that results in death, is life-threatening, requires inpatient hospitalization/prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is medically important.
Maternal Participants With Adverse Event of Special Interest (AESI) | From randomization up to 24 weeks postpartum
  Maternal participants with an AESI will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. AESIs are considered as infections that are severe, hypoalbuminemia, deep vein thrombosis and/or pulmonary embolism, and clinically significant bleeding.
Maternal Participants with TEAE Leading to Discontinuation of Study Intervention | Up to Week 104
  Maternal participants with TEAE leading to discontinuation of study intervention will be reported.
Neonate/Infant with TEAE | Up to Week 104
  Neonatal/infant participants with a TEAE will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Neonate/Infant with SAE | Up to Week 104
  Neonatal/infant participants with SAE will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. An SAE is any untoward medical occurrence that at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is medically Important.
Neonate/Infant with AESI | Up to Week 104
  Neonatal/infant participants with AESI will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. AESIs are considered as: In infants- clinically significant mortalities in fetus/neonates due to maternal infections, and hypogammaglobulinemia.
Fetus/Neonate With TEAE of Bleeding | Up to Week 104
  Fetus/Neonate with TEAE of Bleeding will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. Treatment-emergent AEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Neonate With TEAE of Infection | Up to Week 104
  Neonate with TEAE of Infection will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. Treatment-emergent AEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Infant Development as Measured by Bayley Scales at Week 52 and Week 104 | At Week 52 and 104
  The Bayley Scales of Infant and Toddler Development include a set of individually administered developmental scales designed to measure current developmental functioning in infants and toddlers up to 42 months of age in the areas of cognition, language, motor skills, social-emotional, and adaptive behavior, with age adjusted for prematurity. The cognition, language, motor skills scales are directly administered to the infant, while social-emotional, and adaptive behavior scales are caregiver questionnaires. The scores are standardized using norm reference samples with representative demographics and age adjusted for prematurity.
Maternal Participants With Antibodies to Nipocalimab Including Neutralizing Antibodies in Maternal Serum During Pregnancy and Postpartum | Up to Week 24
  Maternal participants with antibodies to nipocalimab including neutralizing antibodies in maternal serum during pregnancy and postpartum will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Brazil (3):
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- France (2):
  - CHRU Lille, Lille
  - Hopital trousseau- APHP, Paris
- Semmelweis Egyetem, Budapest, Hungary
- Sheba Medical Center, Ramat Gan, Israel
- Italy (2):
  - Mangiagalli Clinic IRCCS Ca Granda Foundation Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Rome
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital HF Ulleval sykehus, Oslo
  - Universitetssykehuset Nord-Norge HF, Tromsø
  - St. Olavs Hospital, Trondheim
- Slovakia (3):
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Univerzitná nemocnica Martin, Martin
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
- Univerzitetni klinicni center Ljubljana, Ljubljana, Slovenia
- Hosp. Virgen Del Rocio, Seville, Spain
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- Centre Hospitalier Universitaire Vaudois CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Tiller H, Tiblad E, Baker P, Van Valkenburgh H, Heerwegh D, Keshinro B. Design of a Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study of Nipocalimab in Pregnancies at Risk for Fetal and Neonatal Alloimmune Thrombocytopenia. Am J Perinatol. 2025 Aug 20. doi: 10.1055/a-2666-5642. Online ahead of print. PMID 40720970